CLINICAL TRIAL: NCT01912209
Title: Baptist Employee Healthy Heart Study (BEHHS) - A Novel Web-based Approach to Reduce Cardiovascular Disease Risk in a Diverse Employee Population With Metabolic Syndrome Via Diet and Lifestyle Change
Brief Title: A Web-based Approach to Treating Cardiovascular Disease Risk in Employees With Metabolic Syndrome
Acronym: BEHHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-028
Record Dates: First submitted 2013-07-03; First posted 2013-07-31 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Metabolic Syndrome; Cardiovascular Disease; Atherosclerosis; Obesity
Keywords: employees; metabolic syndrome; obesity; sub-clinical cardiovascular disease; weight loss; diet
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Atherosclerosis; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- My Everyday Health Group (Experimental): Subjects in this group will be randomized to a web based diet and weight modification program (MyEveryday Health) and provided personal access codes. They will also continue to have access to the WebMD website provided as part of their employment with Baptist Health South Florida.
  Interventions: Behavioral: My Everyday Health
- WebMD Group (No Intervention): This group will continue to have access to a website that is available for use of all employees (WebMD) at Baptist Health South Florida. This is the care-as-usual arm.

INTERVENTIONS:
Behavioral: My Everyday Health — MyEveryday Health is a web-based nutritional and lifestyle management program. The program includes personalized diet and weight guidance, meal planners, shopping list generator, recipe finder, weight tracker and dining out and fast food guides. Based on specific algorithms, tips and suggestions on how to make changes in their diet and lifestyle will be give each time the subject logs in. The MyEverydayHealth website will also be available as an app for their smart phone to the participants. If they choose to use the app, daily reminders to log in and use their tools will be sent, along with motivating tool/tips/tricks to stay with the program.
  Arms: My Everyday Health Group

SUMMARY:
The purpose of BEHHS is first to assess the baseline sub-clinical disease in a population of Baptist Health Employees who have Metabolic Syndrome, a known contributor to cardiovascular disease. Second, the investigators wish to encourage a healthy lifestyle through personalized nutrition and fitness advice, delivered as part of a web based program, which will in turn lead to increases in heart healthy behaviors such as increased consumption of heart healthy foods, increased exercise initiation, and more positive attitudes about health. To assess this, the investigators plan to randomize 200 employees with Metabolic Syndrome to either the new web-based diet and lifestyle program, or to care-as-usual, which is the currently offered MyWellnessAdvantage and WebMD websites. The investigators hypothesize that the web-based group will show greater improvements in physical health (such as weight loss, cholesterol reduction, etc.) as well as increased consumption of heart healthy foods, exercise initiation, and quality of sleep as measured by surveys administered at the 4,8, and 12 month follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Baptist Health
* Access to Internet
* Has a smart phone (Android or Apple supported) with data plan
* Has an email address
* Diagnosis of three or more of the following:

  1. Waist circumference >=40 inches in and male and >= 35 inches in a female
  2. Fasting triglyceride level > 150 mg/dl*
  3. HDL-C < 40 mg/dl in men or < 50 mg/dl in women*
  4. BP > 130/85 mm Hg*
  5. Fasting blood glucose > 110 mg/dl

     * Or currently on medication to treat the abnormal condition

Exclusion Criteria:

1. Prior history of major cardiovascular events (angina, myocardial infarction, prior coronary revascularization
2. Any woman of childbearing potential who is pregnant, breastfeeding/currently lactating, seeking to become pregnant or suspects that she may be pregnant**
3. Active treatment for cancer
4. Known history of a bilateral mastectomy
5. Known history of diabetes (already being treated as high-risk group, would not qualify as having Metabolic Syndrome for purposes of our study)
6. Known history of Chronic Obstructive Pulmonary Disease
7. Currently in atrial fibrillation
8. Known history of hypo-tension
9. Known history of heart failure
10. Known history of aortic valve stenosis
11. Known history of heart block
12. Chest CT scan in the last year
13. Cognitive inability as judged by the interviewer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Reduction in BMI | 4 months, 12 months

SECONDARY OUTCOMES:
Change in waist circumference | 4 months, 12 months
Change in Lipids | 4 months, 12 months
  Examining any changes in advanced lipids such as HDL, LDL, triglycerides, particle size
Change in Blood Pressure | 4 months, 12 months
Change in Glucose Regulation | 4 months, 12 months
  Change in fasting blood glucose(FBG) and HbA1C
Lifestyle Change | 4 months, 12 months
  Changes in reported physical activity, diet, and behavioral scores based on self report by survey
Change in Sub-Clinical Disease | 12 months
  Change in measures of sub-clinical cardiovascular disease; Endothelial function, Carotid intima-medial thickness, coronary artery calcium

CONTACTS AND LOCATIONS:
Overall Officials: Khurram Nasir, MD, MPH, Principal Investigator — Baptist Health Medical Group
Locations (1):
- South Miami Heart Center Outpatient Services, Miami, Florida, United States

REFERENCES:
- [Derived] Aziz M, Gannarapu S, Humayun C, Siddiqui U, Nasir K, Aneni EC. Association of particles of lipoprotein subclasses with arterial stiffness in a high-risk working population: the Baptist Employee Healthy Heart Study (BEHHS). Egypt Heart J. 2020 Mar 19;72(1):12. doi: 10.1186/s43044-020-00046-4. PMID 32193785
- [Derived] Post JM, Ali SS, Roberson LL, Aneni EC, Shaharyar S, Younus A, Jamal O, Ahmad R, Aziz MA, Malik R, Spatz ES, Feldman T, Fialkow J, Veledar E, Cury RC, Agatston AS, Nasir K. Rationale and design of the Baptist Employee Healthy Heart Study: a randomized trial assessing the efficacy of the addition of an interactive, personalized, web-based, lifestyle intervention tool to an existing health information web platform in a high-risk employee population. Trials. 2016 Jul 1;17(1):308. doi: 10.1186/s13063-016-1424-z. PMID 27369488